CLINICAL TRIAL: NCT05825248
Title: Comparing Two Protocols to Improve Reflex Integration and Functional Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Salus University (Other)
Responsible Party: Principal Investigator, Healey Miller, Principal Investigator, Salus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H.Miller.2.27.23
Record Dates: First submitted 2023-03-09; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Developmental Delay
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Intervention Model Description: participants will be assigned to one of two groups. Each group will recieve the same minutes of treatment however one group will include reflex integration and one will include fine and gross motor intervention (standard OT treatment) only.
Who Masked: Outcomes Assessor
Masking Description: Outcome measures will be administered and scored by a masked examiner who is licensed to practice occupational therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reflex integration + fine and gross motor treatment (Experimental): For 20 minutes per week for 8 weeks, this group will recieve 10 minutes of fine and gross motor treatment and 10 minutes of reflex integration exercises from the Move Play Thrive program.
  Interventions: Other: Reflex integration + fine and gross motor treatment
- Fine and gross motor treatment only (Active Comparator): For 20 minutes per week for 8 weeks, this group will recieve 20 minutes of standard occupational therapy treatment consisting of fine and gross motor intervention.
  Interventions: Other: Fine and gross motor treatment only

INTERVENTIONS:
Other: Fine and gross motor treatment only — occupational therapy intervention involving general fine and gross motor activities
  Arms: Fine and gross motor treatment only
Other: Reflex integration + fine and gross motor treatment — occupational therapy intervention involving general fine and gross motor activities as well as targeted reflex integration exercises
  Other Names: Move, Play, Thrive reflex integration exercises
  Arms: Reflex integration + fine and gross motor treatment

SUMMARY:
The goal of this quantitative experimental study is to compare two occupational therapy interventions intended to improve functional skills. The main questions it aims to answer are:

Question 1: Do preschool children who participate in occupational therapy intervention designed to promote integration of the TLR reflex in conjunction with fine and gross motor intervention demonstrate improved integration of the TLR reflex in clinical assessment, compared to children who participate in fine and gross motor intervention only for an equal amount of time?

Question 2: Do preschool children who participate in occupational therapy intervention designed to promote integration of the TLR reflex in conjunction with fine and gross motor intervention demonstrate improved integration of the TLR reflex in clinical assessment, compared to children who participate in fine and gross motor intervention only for an equal amount of time?

Participants will participate in either a therapy program consisting of either fine and gross motor treatment in conjunction with reflex integration treatment, or fine and gross motor treatment only.

If there is a comparison group: Researchers will compare the group recieving reflex integration in conjunction with fine and gross motor treatment and the fine and gross motor only group to see if one is more effective at integrating the reflex and/or improving functional skills.

DETAILED DESCRIPTION:
Pre-intervention, INPP screening for TLR will be administered to determine eligibility for the study and baseline of reflex persistence. the Peabody Developmental Motor Scales 2nd Edition (PDMS2) stationary and visual motor integration sections will be administered to assess fine and gross motor skills. Stratified random sampling will be used to create two parallel groups. Both the INPP and PDMS2 will be administered and scored by a masked examiner who is licensed to practice occupational therapy.

For 6 weeks, one group will receive 20 minutes standard occupational therapy intervention while the second group will receive 10 minutes of standard occupational therapy intervention and 10 minutes of TLR integration protocol (Move Play Thrive Program). 20 minutes per week is standard treatment time for preschool occupational therapy sessions in Aberdeen School District. Intervention will be provided by the PI, Healey Miller.

Post-intervention, the Peabody Developmental Motor Scales 2nd Edition (PDMS2) stationary and visual motor integration sections will be re-administered to assess fine and gross motor skills and the INPP screening for TLR will be re-administered to assess for retained TLR reflex. Both the INPP and PDMS2 will be administered and scored by a masked examiner who is licensed to practice occupational therapy. Data will be reviewed to determine if the progress made between groups, in regard to motor skills and reflex integration, is statistically significant. Data will be reviewed to compare progress made in each group in fine/gross motor skills and reflex integration, and to determine if changes made are statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 3 to <6 years old
* Attending preschool at Hopkins Preschool, Stevens Elementary Preschool, or Central Park Preschool within Aberdeen School District
* Receiving weekly occupational therapy services to address fine motor, gross motor, or sensory deficits
* Displays signs of retained tonic labyrinthine reflex (TLR) after a brief INNP TLR screening test (a score of 3, or 4 will be considered a retained TLR for the purpose of this study)

Exclusion Criteria:

* Students enrolled in an alternative enrollment format
* Students who are absent for a consecutive period of 5 or more school days

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline functional skills at 8 weeks | week 0 and week 8
  functional skills as measured by the Peabody Developmental Motor Scales Stationary and Visual Motor Integration sections. This standardized test scoring can be converted into z-scores for data comparison.
Change from baseline TLR inegration at 9 weeks | week 0 and week 8
  integration of the tonic labyrinthine reflex as measured by the INPP measure for retained primitive reflexes. INPP scale 0-4, 0 being no reflex retained and 4 being severe reflex retention

CONTACTS AND LOCATIONS:
Overall Officials: Healey Miller, Principal Investigator — Salus University
Locations (1):
- Aberdeen School District, Aberdeen, Washington, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers